CLINICAL TRIAL: NCT01147081
Title: A Phase III, Multicenter, Uncontrolled, Open-label Study to Evaluate Safety and Immunogenicity of Begrivac®, Preservative Free, Inactivated Split Influenza Vaccine, Using the Strain Composition 2010/2011 When Administered to Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity, Inactivated Split Influenza Vaccine, Using the Strain Composition 2010/2011
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V44_14S; 2010-018371-18
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Seasonal Influenza
Keywords: Influenza vaccine; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: BEGRIVAC

INTERVENTIONS:
Biological: BEGRIVAC — 126 healthy subjects enrolled to receive, in open-label manner, one dose of Begrivax (influenza vaccine)

SUMMARY:
Annual trial for registration influenza vaccine Begrivac with strain composition for season 2010/2011.

DETAILED DESCRIPTION:
At enrolment, subjects were stratified into two age strata (18 to 60 years, over 60 years). Total duration of the study is three weeks. Vaccinations were to be administered on day 1. Blood samples were collected at day 1 (baseline, before the vaccination) and at day 22 (three weeks after the vaccination). Sera were tested by Hemagglutination Inhibition (HI) assay. Safety was assessed until 3 weeks after the vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers of 18 years of age and older, mentally competent, willing and able to give written informed consent prior to study entry;
2. Individuals able to comply with all the study requirements;
3. Individuals in good health as determined by medical history, physical examination and clinical judgment of the investigator.

Written informed consent must be obtained for all the subjects before enrollment into the study after the nature of the study has been explained.

Exclusion Criteria:

1. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study;
2. Individuals with any serious chronic or acute disease (in the judgment of the investigator), including but not limited to:

   1. Cancer, except for localized skin cancer;
   2. Advanced congestive heart failure;
   3. Chronic obstructive pulmonary disease (COPD);
   4. Autoimmune disease (including rheumatoid arthritis);
   5. Acute or progressive hepatic disease;
   6. Acute or progressive renal disease;
   7. Severe neurological or psychiatric disorder;
   8. Severe asthma;
3. Individuals with history of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g. to ovalbumin, chicken protein, chicken feathers, influenza viral protein, Polymyxin B;
4. Individuals with known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting, for example, from:

   1. receipt of immunosuppressive therapy (any parenteral or oral corticosteroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study;
   2. receipt of immunostimulants;
   3. receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study;
   4. suspected or known HIV infection or HIV-related disease;
5. Individuals with known or suspected history of drug or alcohol abuse;
6. Individuals with a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject;
7. Female who are pregnant or nursing (breastfeeding) mothers or females of childbearing age do not plan to use acceptable birth control measures, for the duration of the study. Adequate contraception is defined as hormonal (e.g., oral, injection, transdermal patch, implant, cervical ring), barrier (e.g., condom with spermicide or diaphragm with spermicide),,intrauterine device (IUD), or monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject's study entry;
8. Individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study;
9. Individuals that within the past 12 months have received more than one injection of influenza vaccine;
10. Individuals that within the past 6 months have:

    1. had laboratory confirmed seasonal or pandemic influenza disease;
    2. received seasonal or pandemic influenza vaccine;
11. Individuals with any acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days
12. Individuals that have experienced fever (i.e., axillary temperature ≥ 38°C) within the last 3 days of intended study vaccination
13. Individuals participating in any clinical trial with another investigational product 4 weeks prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.
14. Individuals who received any other vaccines within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccines
15. Individuals who have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks and for the full length of the study
16. Individuals who are part of study personnel or close family members conducting this study.
17. Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.
18. BMI > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of antibody response to each influenza vaccine antigen, as measured by haemagglutination inhibition (HI) test on Day 1 and on Day 22, and evaluation of safety of Begrivac | 22 days (-1/+5)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- Germany (3):
  - Hamburg, Hamburg
  - Universität Rostock/Medizinische Fakultät, Ernst-Heydemann Str. 6, Rostock
  - Magdeburg, Saxony-Anhalt

REFERENCES:
- [Derived] Loebermann M, Anders G, Brestrich G, Fritzsche C, Klammt S, Borso D, Frimmel S, Riebold D, Reisinger EC. Safety and immunogenicity of a trivalent single dose seasonal influenza vaccine containing pandemic A(H1N1) antigen in younger and elderly subjects: a phase III open-label single-arm study. Vaccine. 2011 Feb 1;29(6):1228-34. doi: 10.1016/j.vaccine.2010.11.092. Epub 2010 Dec 15. PMID 21167116